CLINICAL TRIAL: NCT04863625
Title: Effects of a Peer-led Educational Intervention Based on Theory of Planned Behavior on Substance Use Intentions and Behaviors Among Secondary School Students of Dessie and Kombolcha Town, Northeast Ethiopia: a Quasi- Experimental Study
Brief Title: Effects of a Peer-led Educational Intervention Based on Theory of Planned Behavior on Substance Use Intentions and Behaviors Among Secondary School Students of Dessie and Kombolcha Town, Northeast Ethiopia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wollo University (Other)
Collaborators: Jimma University (Other)
Responsible Party: Principal Investigator, Yitbarek Wasihun, EEffects of a peer-led educational intervention based on theory of planned behavior on substance use intentions and behaviors among secondary school students of dessie and kombolcha town, northeast Ethiopia: a quasi- experimental study, Wollo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021
Record Dates: First submitted 2021-04-26; First posted 2021-04-28 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Substance Use
Keywords: Substance use, alcohol ,cigarette and Khat
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The intervention will be a peer education process on substance use (smoking, drinking and chewing) prevention based on the Theory of Planned Behavior (TPB). This program is a Level I, primary prevention; thus, it is an early intervention program. The program is targeting students with all substance experience (non-user, current user, and ever users).
  The intervention aims to encourage anti-substance attitudes and beliefs; foster perceptions of normative support for anti-substance behavior; increase perceptions of control/self-efficacy to resist substance use, increase knowledge and risk perceptions on substance and decrease in intention to use substance and actual substance use behaviors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 748 students from two secondary schools for the intervention group will be selected and participated in a peer led education process on substance use (smoking, drinking and chewing) prevention based on the Theory of Planned Behavior (TPB).
  Interventions: Behavioral: a peer-led educational intervention based on theory of planned behavior on substance use intentions and behaviors
- Control group (No Intervention): 748 students from two secondary schools for the control group will selected and receive t their school's regular curriculum.

INTERVENTIONS:
Behavioral: a peer-led educational intervention based on theory of planned behavior on substance use intentions and behaviors — The intervention will be a peer led education process on substance use (smoking, drinking and chewing) prevention based on the Theory of Planned Behavior (TPB).The intervention aims to encourage anti-substance attitudes and beliefs; foster perceptions of normative support for anti-substance behavior; increase perceptions of control/self-efficacy to resist substance use, increase knowledge and risk perceptions on substance and decrease in intention to use substance and actual substance use behaviors. Six education sessions will be delivered, with one session occurring each week. Each session will be lasted 40-55 minutes. The intervention will be conducted in 30 groups of selected students from grade 9-12, a pair of peer educators will educate a 30 sized group weekly (30 students /group)/ classrooms at pre-assigned time during class periods. The six sessions will be guided by four student training modules.
  Arms: Experimental group

SUMMARY:
This study aims to measure the effects of a per-led educational intervention based on theory of planned behavior to reduce tobacco, alcohol and khat use and intention to use among secondary school students over 3-months of follow-up in Dessie and Kombolcha town, Northeast Ethiopia.

DETAILED DESCRIPTION:
This study aims to measure the effects of a per-led educational intervention based on theory of planned behavior to reduce tobacco, alcohol and khat use and intention to use among secondary school students over 3-months of follow-up in Dessie and Kombolcha town, Northeast Ethiopia.A quasi-experimental nonequivalent control group pretest-post-test design will be carried out among secondary school students of Dessie and Kombolcha Town from April to August, 2021. Individuals/Students/ in those selected schools will be allocated as intervention and control group purposively. The study will include 748 students from two secondary schools for the intervention group and another 748 students for the control group from other two secondary schools. The per-educational intervention will be planned based on results of the elicitation and TPB constructs and will be implemented on the experimental group for three months. Both experimental and control groups will be followed up after three months of educational intervention using the same tools and methods on same participants interviewed in pretest survey. Primary outcomes are substance(Cigarette,alcohol and Khat) use intention and behavior. Secondary outcome are attitudes, subjective norms, and perceived behavioral control over substance(Cigarette,alcohol and Khat) use. Self-administered questionnaire based on TPB constructs will be used to collect the baseline and follow up data. In-depth interviews will be employed to explore the salient beliefs about substance use. The data will be analyzed using SPSS statistical software package version 20 using appropriate statistical tests including paired t-test, independent t-tests, McNemar and multivariate logistic regression analysis. All statistical tests will be carried out using two tailed tests with alpha set at 0.05. Information from the interviews will be transcribed verbatim, analyzed, and coded thematically.

ELIGIBILITY:
Inclusion Criteria:

* All Grade 9-12 students, both girls and boys with any substance use experience (non-user, current user, and ever users) (aged 15-24 years) attending the four secondary schools of Dessie and Kombolcha town are eligible.

Exclusion Criteria:

* Grade 9-12 students who are not wanting to attend the evaluation and not able to have a follow- up will be excluded from the study.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1496 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Behavioral Intention to smoke cigarette over a 3-month period | Three months
  It is the secondary school student motivation in the sense of his/her conscious plan to exert such behavior, intent to use cigarette. It will be assessed by a 3-item self-report questionnaire designed for the study, based on the manual for constructing questionnaires based on the TPB (Francis, et al. 2004). Participants could score between 3 -21, with a low score indicating no intention to use tobacco, over a 3-month period and a high score indicating an intention to use tobacco over a 3-month periods.
Behavioral Intention to drink alcohol over a 3-month period | Three months
  It is the secondary school student motivation in the sense of his/her conscious plan to exert such behavior, intent to use alcohol. It will be assessed by a 3-item self- report questionnaire designed for the study, based on the manual for constructing questionnaires based on the TPB (Francis, et al. 2004). Participants could score between 3 -21, with a low score indicating no intention to use alcohol, over a 3-month period and a high score indicating an intention to use alcohol over a 3-month periods.
Behavioral Intention to chew khat over a 3-month period | Three months
  It is the secondary school student motivation in the sense of his/her conscious plan to exert such behavior, intent to use khat. It will be assessed by a 3-item self-report questionnaire designed for the study, based on the manual for constructing questionnaires based on the TPB (Francis, et al. 2004). Participants could score between 3 -21, with a low score indicating no intention to use khat, over a 3-month period and a high score indicating an intention to use khat over a 3-month periods

CONTACTS AND LOCATIONS:
Locations (1):
- Wollo University, Dessie, Addise Abeba, Ethiopia

IPD SHARING:
Plan to Share IPD: No
All individual participant data will be available to other researchers during and after publication